CLINICAL TRIAL: NCT05085626
Title: An Open, Multi-center, Cohort Clinical Study of Fluzoparib in Combination With Chidamide or Camrelizumab for HRD Positive and HER2-negative Advanced Breast Cancer
Brief Title: Fluzoparib in Combination With Chidamide or Camrelizumab for HRD Positive HER2 Negative Advanced Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BC-Fluzoparib
Record Dates: First submitted 2021-06-29; First posted 2021-10-20 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Advanced HER2 Negative Breast Carcinoma; HRD+Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fluzoparib+chidamide (Experimental): Fluzoparib: 150 mg twice daily (morning and evening) for 21 consecutive days as a cycle until disease progression or intolerance.
  Chidamide: It is recommended to take 20 mg (4 tablets) twice a week, with an interval of no less than 3 days between doses (such as Monday and Thursday, Tuesday and Friday, Wednesday and Saturday, etc.), for 30 minutes. Until disease progression or intolerable to patient.
  Interventions: Drug: fluzoparib+chidamide
- fluzoparib+camrelizumab (Experimental): Fluzoparib: 150 mg twice daily (morning and evening) for 21 consecutive days as a cycle until disease progression or intolerance.
  Camrelizumab: 200 mg IV drip over approximately 30 minutes (no less than 20 minutes and no more than 60 minutes) on Day 1 of each 3-week treatment cycle until disease progression or intolerance.
  Interventions: Drug: fluzoparib+camrelizumab

INTERVENTIONS:
Drug: fluzoparib+chidamide — Arms A will be treated with fluzoparib in combination with cedaramide
  Arms: fluzoparib+chidamide
Drug: fluzoparib+camrelizumab — Arms B will be treated with fluzoparib in combination with camrelizumab
  Arms: fluzoparib+camrelizumab

SUMMARY:
This study is planned to include 40 patients with HER2-negative advanced breast cancer to receive fluzoparib combined with chidamide or fluzoparib combined with camrelizumab to observe and evaluate the efficacy and safety of fluzoparib combined with camrelizumab or chidamide in the treatment of HRD-positive HER2-negative advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. histologically confirmed initial stage IV breast cancer or recurrent metastatic breast cancer; advanced treatment stage received at least 1 line of chemotherapy but no more than 2 lines of chemotherapy; hormone receptor-positive patients received at least one endocrine therapy in advanced treatment stage, or the investigator judged that they were not suitable for endocrine therapy; and patients with hormone receptor-positive advanced breast cancer who progressed within 2 years of adjuvant endocrine therapy.
2. histologically confirmed invasive HER2-negative breast cancer (specific definition: HER20-1 + or HER2 2 + by immunohistochemistry but negative or no amplification by FISH or CISH, following the 2018 version of the ASCO-CAPHER2 guidelines for negative interpretation);
3. central confirmation of HRD positivity, known germline BRCA and/or systemic BRCA mutation status is allowed to be preferred.
4. age 18-70 years
5. According to RECIST 1.1, at least one measurable lesion is present;
6. ECOG score: 0-2; expected survival more than 12 weeks;
7. Previous treatment with immune checkpoint inhibitors, PARP inhibitors and HDAC inhibitors (including chidamine, romidepsin, vorinostat, benirestat, parastat, etc.);
8. All acute toxicities caused by previous anti-tumor treatment return to the level specified in the inclusion/exclusion criteria (except alopecia and other toxicities that are considered by the investigator to pose no safety risk to the subjects);
9. Female subjects of childbearing potential need to use a medically recognized contraceptive measure during the study treatment and at least 3 months after the last use of the study drug;
10. Patients with known hormone receptor status;
11. Main organ function is basically normal, and meet the following conditions:

    1. Blood routine examination criteria need to meet: HB ≥ 90 g/L (14 without blood transfusion); ANC ≥ 1.5 × 109/L; PLT ≥ 75 × 109/L;
    2. Biochemical examination need to meet the following criteria: TBIL ≤ 1.5 × ULN (upper limit of normal); ALT and AST ≤ 3 × ULN; if there is liver metastasis, ALT and AST ≤ 5 × ULN; serum Cr ≤ 1 × ULN;
    3. cardiac function: LVEF ≥ 50%
12. The subject voluntarily joined the study and signed the informed consent form.

Exclusion Criteria:

1. Uncontrolled central nervous system metastasis (defined as symptoms or requiring glucocorticoids or mannitol to control symptoms);
2. Clinically symptomatic third space effusion, pericardial effusion, pleural effusion and abdominal effusion that cannot be controlled by pumping or other treatments;
3. Currently or recently (within 30 days before enrollment) is participating in another clinical study;
4. Five Other malignant tumors (except adequately treated cervical carcinoma in situ or skin squamous cell carcinoma or controlled skin basal cell carcinoma) within the past 4 years;
5. Uncontrolled cardiac clinical symptoms or diseases, such as: (1) NYHA grade 2 or higher heart failure (2) unstable angina pectoris (3) myocardial infarction within 1 year (4) clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention (5) QTc > 470 ms;
6. Hyperactive/venous thrombotic events, such as cerebrovascular accidents (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep venous thrombosis and pulmonary embolism;
7. He following history 24 days before signing the ICF: gastrointestinal ulcers, gastrointestinal perforation, corrosive esophagitis or gastritis, inflammatory bowel disease or inflammation, abdominal fistula, tracheoesophageal fistula or intra-abdominal abscess;
8. Factors that significantly affect oral drug absorption, such as inability to swallow, chronic diarrhea and intestinal obstruction;
9. Patients with a clear history of allergy, Potential allergy or intolerance to cidaniline, fluzoparib, and carreizumab;
10. Human immunodeficiency virus (HIV) infection, active hepatitis B (hepatitis B surface antigen positive and HBV DNA ≥ 500 IU/ml), hepatitis C (hepatitis C antibody positive and HCV-RNA above the lower limit of detection of the analytical method);
11. Female patients during pregnancy and lactation, female patients of childbearing potential with positive baseline pregnancy test or female patients of childbearing age who are unwilling to take effective contraceptive measures throughout the trial;
12. According to the investigator's judgment, the presence of concomitant diseases (including but not limited to hypertension with poor drug control, severe diabetes, neurological or psychiatric diseases, active infection, etc.) or any other condition that seriously endangers the subject's safety, may confound the study results, or affect the subject's completion of this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-02-08 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR(objective response rate) | At the end of Cycle 1 (each cycle is 28 days)
  through study completion, an average of 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No